CLINICAL TRIAL: NCT04533022
Title: A Phase 2, Multi-Centre, Open-Label, Single-Arm Trial Investigating the Safety, Efficacy and Pharmacokinetics of C21 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Safety, Efficacy and Pharmacokinetics of C21 in Subjects With IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vicore Pharma AB (Industry)
Collaborators: Orphan Reach Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-C21-005; 2020-000822-24 (EudraCT Number)
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — compound 21

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C21 (Experimental): C21 100 mg BID (twice daily)
  Interventions: Drug: C21

INTERVENTIONS:
Drug: C21 — C21 100 mg BID (twice daily)
  Other Names: Buloxibutid, Compound 21

SUMMARY:
This trial is a multi-centre, open-label, single-arm phase 2 trial investigating the safety, efficacy and pharmacokinetics of C21 in subjects with idiopathic pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, consistent with ICH-GCP R2 and local laws, obtained before the initiation of any trial related procedure
2. A diagnosis of IPF within 5 years prior to Visit 1, as per either ATS/ERS/JRS/ATLAT/Fleischner guidelines
3. Age ≥40 years
4. Forced vital capacity (FVC) ≥60% predicted at Visit 1 (specifically for UK: FVC ≥80% predicted at Visit 1)
5. Forced expiratory volume in the first sec (FEV1)/FVC ratio ≥0.7 prebronchodilator at Visit 1
6. Oxygen saturation (SpO2) >85% by pulse oximetry while breathing ambient air at rest at Visit 1
7. High-resolution computed tomography (HRCT) within 36 months prior to Visit 1 with central reading demonstrating either a or b, and c:

   a. A pattern consistent with usual interstitial pneumonitis (UIP) according to ATS/ERS/JRS/ALAT or Fleischner guidelines i. UIP ii. Probable UIP or b. A pattern indeterminate for UIP according to either ATS/ERS/JRS/ALAT or Fleischner guidelines and a historical biopsy consistent with IPF c. Extent of fibrosis > extent of emphysema
8. Fully vaccinated against COVID-19 prior to screening (Visit 1). Subjects are considered fully vaccinated for COVID-19 ≥14 days after they have received vaccination dose(s) according to local label

Exclusion Criteria:

1. Previous use of antifibrotic treatment for an interstitial lung disease (e.g. nintedanib or pirfenidone) for > 6 months
2. Smoking (including e-cigarettes) within 6 months prior to Visit 1
3. Body mass index (BMI) >35 or <18
4. IPF exacerbation within 3 months prior to Visit 1:

   * Acute worsening or development of dyspnoea typically <1 month duration
   * Computed tomography with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia pattern (if no previous computed tomography is available, the qualifier "new" can be dropped)
   * Deterioration not fully explained by cardiac failure or fluid overload
5. Concurrent serious medical condition with special attention to cardiac or ophthalmic conditions (e.g. contraindications to cataract surgery) which in the opinion of the investigator makes the subject inappropriate for this trial
6. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma and cervical intraepithelial neoplasia grade I
7. Treatment with any of the medications listed below within 4 weeks prior to Visit 1:

   * Cytochrome p450 (CYP) 3A4 inducers (e.g. rifampicin, phenytoin, St. John's Wort)
   * CYP3A4 inhibitors (e.g. clarithromycin, ketoconazole, nefazodone, itraconazole, ritonavir)
   * Medicines that are substrates of CYP1A2, CYP3A4 or CYP2C9 with a narrow therapeutic range
   * Experimental drugs
   * Any systemic immunosuppressive therapies other than:
   * Inhaled corticosteroids which can be used throughout the trial period provided the dose is kept stable
   * Corticosteroids for the treatment of acute exacerbations
   * The continuation of stable doses of ≤15 mg daily doses of prednisolone
8. Treatment with any of the medications listed below within 2 weeks prior to Visit 1:

   * Proton pump inhibitors (PPI's) more than once daily
   * Histamine H2 receptor antagonists (H2RA's)
   * Sulphasalazine and rosuvastatin
   * High dose breast cancer resistance protein sensitive substrates (other than sulphasalazine or rosuvastatin)
9. Any of the following findings at Visit 1:

   * Prolonged QTcF (QT interval with Fridericia's correction) (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG, as judged by the Investigator
   * Positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCVAb) or human immunodeficiency virus 1+2 antigen/antibody (HIV 1+2 Ag/Ab)
   * Positive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin)
10. Inability to generate lung function data at Visit 1 meeting the minimum standards of the ATS/ERS 2005 guideline, as determined by central review
11. Clinically significant abnormal laboratory value at Visit 1 indicating a potential risk for the subject if enrolled in the trial as evaluated by the investigator
12. Pregnant or breast-feeding female subjects
13. Female subjects of childbearing potential not willing to use contraceptive methods
14. Male subjects not willing to use contraceptive methods
15. Subjects not willing to adhere to dietary restrictions during the trial period
16. Participation in any other interventional trial during the trial period
17. Subjects known or suspected of not being able to comply with this trial protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
18. Discontinuation or change of previous antifibrotic treatment (e.g. nintedanib or pirfenidone) due to disease progression

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Porter, MD, Principal Investigator — Respiratory Medicine, University College Hospital
Locations (21):
- India (11):
  - AMCMET Medical College and Sheth LG General Hospital, Ahmedabad, Gujarat
  - Unity Hospital, Surat, Gujarat
  - The Bhatia Hospital, Mumbai, Maharashtra
  - Grant Government Medical Collage and Sir J.J. Group of Hospitals, Mumbai, Maharashtra
  - N. K. P. Salve Institute of Medical Sciences & Research Centre and Lata Mangeshkar Hospital, Nagpur, Maharashtra
  - Ace Hospital & Research Center, Pune, Maharashtra
  - Oyster & Pearl Hospitals, Pune, Maharashtra
  - Hindusthan Hospital, Coimbatore, Tamil Nadu
  - Jawaharlal Nehru Medical College - Aligarh Muslim University, Aligarh, Uttar Pradesh
  - Midland Healthcare and Research Centre, Lucknow, Uttar Pradesh
  - Apollo Spectra Hospitals (Apollo Speciality Hospital Pvt. Ltd.), Kanpur
- Clinical Hospital for Emergency Medical Care n.a. N.V. Solovyev, Yaroslavl, Russia
- Ukraine (4):
  - MNCE City Clinical Hospital, Kharkiv
  - Lviv National Medical University, Lviv
  - Odessa Regional Hospital, Odesa
  - Private Small Scale Enterprise Medical Center 'PULSE', Vinnytsia
- United Kingdom (5):
  - University Hospital Birmingham, Birmingham
  - Royal Brompton Hospital, London
  - University College Hospital, London
  - University College London Hospitals, London
  - Medicines Evaluation Unit, Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 participants were enrolled and received at least one dose of C21. 138 participants signed informed content and were screened, however, 86 of those were screening failures and thus not enrolled.
Groups:
- C21 100 mg BID: Oral administration of 100 mg BID C21 (200 mg daily)
Period: Overall Study
Arm/Group | C21 100 mg BID
Started | 52
Completed | 27
Not Completed | 25
Not completed — Withdrawal by Subject | 15
Not completed — Adverse Event | 6
Not completed — Death | 1
Not completed — FVC decline and FVCpp<60% | 2
Not completed — FVC decline, FVCpp<60% and worsening of respiratory symptoms | 1

BASELINE CHARACTERISTICS:
Groups:
- C21 100 mg BID, SAS: Oral administration of 100 mg BID C21 (200 mg daily) Safety analysis set (SAS)
Arm/Group | C21 100 mg BID, SAS
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.3 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 52
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Ukraine | 4
  United Kingdom | 7
  India | 38
  Russia | 3
Height [Mean (Standard Deviation); unit: cm] | 161.69 (8.723)
Weight [Mean (Standard Deviation); unit: kg] | 64.64 (14.178)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 24.57 (4.119)
Smoking status [Count of Participants; unit: Participants]
  Current | 0
  Former | 10
  Never | 42
  Missing | 0
E-cigarettes and vapes status [Count of Participants; unit: Participants]
  Current | 0
  Former | 1
  Never | 51
  Missing | 0
Time since diagnosis of idiopathic pulmonary fibrosis [Mean (Standard Deviation); unit: Years] | 1.01 (1.195)
Oxygen saturation at screening [Mean (Standard Deviation); unit: Percentage of oxygen saturation] | 95.3 (2.40)
FEV1 [Mean (Standard Deviation); unit: L] — Forced expiratory volume in the first sec
  L | 1.912 (0.528)
FVC [Mean (Standard Deviation); unit: L] — Forced vital capacity
  L | 2.387 (0.667)
FEV1/FVC [Mean (Standard Deviation); unit: ratio] | 0.804 (0.067)
FEV1 (% predicted normal) [Mean (Standard Deviation); unit: Percentage of predicted normal FEV1] | 77.51 (14.687)
FVC (% predicted normal) [Mean (Standard Deviation); unit: Percentage of predicted normal FVC] | 75.46 (13.662)
Age of High-resolution computed tomography (HRCT) scan [Mean (Standard Deviation); unit: Months] | 5.58 (8.720)
Previous use of antifibrotics [Count of Participants; unit: Participants]
  Nintedanib | 0
  Pirfenidone | 0
HRCT pattern (central reading) [Count of Participants; unit: Participants] — A high-resolution computed tomography (HRCT) within 36 months prior to Visit 1 was obtained and the pattern categorized.
  Participants
    Typical usual interstitial pneumonitis (UIP) HRCT Pattern | 20
    Probable UIP HRCT Pattern | 32
    HRCT Feature most consistent with Non-IPF diagnosis | 0
    Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Occurring Over the Trial Period
Description: Number of participants with adverse events occurring over the trial period incl. number of participants with any TEAE, serious TEAEs, TEAEs leading to withdrawal from trial, TEAEs leading to discontinuation of treatment, treatment-related TEAEs leading to discontinuation of treatment, TEAEs leading to death, and serious treatment-related TEAEs.
  Adverse events were recorded from signing of informed consent until end of trial.
  Nature and frequency of adverse events are presented in details in the adverse events section.
Time Frame: Trial period of 36 weeks
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | C21 100 mg BID, SAS
Number analyzed (Participants) | 52
Participants
  Total number of subjects with treatment-emergent adverse events (TEAEs) | 37
  Total number of subjects with serious TEAEs | 5
  Total number of subjects with TEAEs leading to withdrawal from study | 6
  Total number of subjects with TEAEs leading to discontinuation of treatment | 12
  Total number of subjects with treatment-related TEAEs leading to discontinuation of treatment | 3
  Total number of subjects with TEAEs leading to death | 2
  Total number of subjects with serious treatment-related TEAEs | 0

2. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Non-imputed Data)
Description: Mean changes in forced vital capacity (FVC) (mL) from baseline to week 12, week 24, and week 36 were calculated
Time Frame: 12, 24, and 36 weeks
Population: Participants in the Full analysis set (FAS) with a measurement.
Measure: Mean (90% Confidence Interval); unit: mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 35
mL
  Week 12 | -4.9 [-73.2 to 63.4]
  Week 24 | 16.0 [-117.4 to 149.3]
  Week 36 | 216.0 [36.9 to 395.1]

3. Secondary Outcome: Change From Baseline in Forced Vital Capacity (Imputed Data)
Description: Mean changes in forced vital capacity (FVC) (mL) from baseline to week 12, week 24, and week 36 were calculated
Time Frame: 12, 24, and 36 weeks
Population: Full analysis set with imputed data
Measure: Mean (90% Confidence Interval); unit: mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 48
mL
  Week 12 | -57.6 [-123.3 to 8.1]
  Week 24 | -70.3 [-170.5 to 29.9]
  Week 36 | 9.4 [-115.6 to 134.4]

4. Secondary Outcome: Rate of Forced Vital Capacity Decline Over Time, FAS
Description: Model-based mean (90% CI) FVC changes over 12, 24, and 36 weeks were normalized to change over 24 weeks.
  A piece-wise linear regression model with knots at weeks 6 and 24 and unstructured covariance matrix was fitted to change from baseline data. Knot selection was performed by visual inspection.
  The model based change over 12, 24, and 36 weeks was normalized to represent a change over 24 weeks.
  Rate of decline was computed as y(t) - y(0) = t*Beta1 + max(0, t-6)*Beta2 + max(0,t-24)*Beta3, adjusted to show the decline per 24 weeks, where y is the value at the respective week and Beta is the model coefficient.
  No imputation of data was conducted.
Time Frame: 12, 24, and 36 weeks
Population: Full analysis set
Measure: Mean (90% Confidence Interval); unit: mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 50
mL
  Week 12 | -8.2 [-141.9 to 125.5]
  Week 24 | 36.4 [-87.1 to 160]
  Week 36 | 108.9 [-4.8 to 222.6]

5. Secondary Outcome: Plasma Concentration of C21 Evaluated in a Sub-set of Subjects, Day 1
Description: The plasma concentration of C21 (ng/mL) was calculated in a subset of subjects at specified timepoints post-dose.
Time Frame: Prior to dosing, 30 min post dose, 1 h post dose, 2 h post dose, 3 h post dose, and 4 h post dose on Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 12
ng/mL
  Prior to dosing | 5.00 (0.00)
  30 min post dose | 1622.0 (1453.64)
  1 h post dose | 1788.11 (1112.48)
  2 h post dose | 864.46 (1062.15)
  3 h post dose | 322.19 (407.29)
  4 h post dose | 282.82 (379.31)

6. Secondary Outcome: Plasma Concentration of C21 Evaluated in a Sub-set of Subjects, Week 12
Description: The plasma concentration of C21 (ng/mL) was calculated at specified timepoints post-dose after 12 weeks of dosing.
Time Frame: Prior to dosing, 30 min post dose, 1 h post dose, 2 h post dose, 3 h post dose, and 4 h post dose at Week 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 8
ng/mL
  Prior to dosing | 27.13 (62.58)
  30 min post dose | 974.28 (1028.90)
  1 h post dose | 1044.02 (1128.30)
  2 h post dose | 794.02 (774.34)
  3 h post dose | 491.25 (820.36)
  4 h post dose | 101.50 (113.96)

7. Secondary Outcome: Plasma Concentration of C21 Evaluated in a Sub-set of Subjects, Week 24
Description: The plasma concentration of C21 (ng/mL) was calculated at specified timepoints post-dose after 24 weeks of dosing.
Time Frame: Prior to dosing, 30 min post dose, 1 h post dose, 2 h post dose, 3 h post dose, and 4 h post dose at Week 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 9
ng/mL
  Prior to dosing | 20.14 (28.608)
  30 min post dose | 615.53 (792.908)
  1 h post dose | 898.61 (779.723)
  2 h post dose | 404.80 (296.002)
  3 h post dose | 151.30 (125.292)
  4 h post dose | 115.93 (151.833)

8. Secondary Outcome: Plasma Concentration of C21 Evaluated in a Sub-set of Subjects, Week 36
Description: The plasma concentration of C21 (ng/mL) was calculated at specified timepoints post-dose after 36 weeks of dosing.
Time Frame: Prior to dosing, 30 min post dose, 1 h post dose, 2 h post dose, 3 h post dose, and 4 h post dose at Week 36
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 9
ng/mL
  Prior to dosing | 89.78 (176.452)
  30 min post dose | 796.29 (839.353)
  1 h post dose | 713.86 (453.540)
  2 h post dose | 298.29 (299.235)
  3 h post dose | 374.16 (459.545)
  4 h post dose | 348.11 (479.786)

9. Secondary Outcome: Cmax in a Sub-set of Subjects
Description: The maximal plasma concentration (Cmax (ng/ml)) was calculated in a subset of subjects after 0, 12, 24, and 36 weeks of dosing
Time Frame: Prior to dosing, 30 min post dose, 1 h post dose, 2 h post dose, 3 h post dose, and 4 h post dose at Weeks 0, 12, 24, and 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 12
ng/mL
  0 Weeks | 1852.13 (80.1)
  12 Weeks | 954.29 (127.9)
  24 Weeks | 524.79 (281.6)
  36 Weeks | 961.86 (73.3)

10. Secondary Outcome: Tmax in a Sub-set of Subjects
Description: The time for the maximal plasma concentration (Tmax (h)) was calculated in a subset of subjects after 0, 12, 24, and 36 weeks of dosing
Time Frame: as for outcome 9
Measure: Median (Full Range); unit: h
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 12
h
  Week 0 | 1.00 [0.5 to 4.0]
  Week 12 | 1.50 [0.5 to 4.0]
  Week 24 | 1.00 [0.0 to 1.0]
  Week 36 | 1.00 [0.5 to 4.00]

11. Secondary Outcome: AUClast in a Sub-set of Subjects
Description: Area under the plasma concentration time curve to the last quantified concentration (AUClast) (h*ng/mL) was calculated in a subset of subjects after 0, 12, 24, and 36 weeks of dosing
Time Frame: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 12
h*ng/mL
  Week 0 | 3018.151 (60.5)
  Week 12 | 1704.924 (126.6)
  Week 24 | 995.600 (213.2)
  Week 36 | 1622.774 (49.8)

12. Secondary Outcome: Accumulation Ratio AUC in a Sub-set of Subjects
Description: Accumulation ratio AUC was calculated in a subset of subjects after 0, 12, 24, and 36 weeks of dosing
Time Frame: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | C21 100 mg BID
Number analyzed (Participants) | 12
Ratio
  Week 12 | 0.84598 (120.5)
  Week 24 | 0.45256 (328.9)
  Week 36 | 0.73765 (67.9)

ADVERSE EVENTS:
Time Frame: Throughout the trial from signing of informed consent until the end-of-trial visit, up to 44 weeks
Description: At each visit the subject was asked about AEs in an objective manner, e.g.: "Have you experienced any problems since the last visit?"
Arm/Group | C21 100 mg BID
All-Cause Mortality (participants affected / at risk) | 2/52
Serious Adverse Events (participants affected / at risk) | 5/52
Other Adverse Events (participants affected / at risk) | 35/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 100 mg BID (N=52)
Angina pectoris (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Sepsis (Cardiac disorders) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | C21 100 mg BID (N=52)
Alopecia (Skin and subcutaneous tissue disorders) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 4 (6)
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (6)
Nausea (Gastrointestinal disorders) | 2 (2)
Blood creatinine increased (Investigations) | 4 (4)
C-reactive protein increased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood glucose increased (Investigations) | 2 (2)
Alanine aminotransferase abnormal (Investigations) | 1 (3)
Aspartate aminotransferase abnormal (Investigations) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (6)
Bundle branch block left (Cardiac disorders) | 3 (3)
Pyrexia (General disorders) | 4 (4)
Influenza like illness (General disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (8)
Lethargy (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT04533022/Prot_SAP_000.pdf